CLINICAL TRIAL: NCT04280991
Title: Exercise During Mild Hypoxia Exposure to Reverse Impaired Glucose Metabolism in Overweight and Obese Humans
Brief Title: Hypoxic Exercise and Glucose Metabolism
Acronym: HYTRIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NL68218.068.18 / METC 18-059
Record Dates: First submitted 2019-07-16; First posted 2020-02-21 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Obesity; Insulin Resistance; Impaired Glucose Tolerance in Obese
Keywords: Metabolism; Hypoxia; Glucose metabolism
MeSH Terms: conditions — Obesity; Insulin Resistance; Hypoxia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate intensity exercise under mild normobaric hypoxia (Experimental): The participants will perform moderate intensity exercise at heart rate corresponding with 50%WMAX (determined during maximal workload test) under mild normobaric hypoxia (FiO2: 15%), two times 30 minutes per day for 4 consecutive days on a cycle ergometer. 24h glucose concentration will be monitored continuously. Afterwards, a meal test challenge will be performed at day 5 to determine fasting/postprandial substrate oxidation.
  Interventions: Other: Moderate intensity exercise under mild normobaric hypoxia and normoxia
- Moderate intensity exercise under normoxia (Placebo Comparator): The participants will perform moderate intensity exercise at 50% WMAX (determined during maximal workload test) under normoxia (FiO2: 21%) two times 30 minutes per day for 4 consecutive days on a cycle ergometer. 24h glucose concentration will be monitored continuously. Afterwards, a meal test challenge test will be performed at day 5 to determine fasting/postprandial substrate oxidation.
  Interventions: Other: Moderate intensity exercise under mild normobaric hypoxia and normoxia

INTERVENTIONS:
Other: Moderate intensity exercise under mild normobaric hypoxia and normoxia — The participant will perform the exercise interventions consisting of cycling at the heart rate corresponding with 50%WMAX (normoxia) or heart rate corresponding with 50% WMAX (hypoxia) for 30 minutes, twice a day, for 4 consecutive days. 24h glucose concentration will be monitored continuously.

SUMMARY:
The obesity epidemic calls for new therapeutic opportunities to prevent and treat obesity and its comorbidities amongst which are insulin resistance and cardiovascular diseases. Recent evidence suggests that tissue oxygenation plays an important role in cardiometabolic health. Remarkably, individuals residing at high altitude (hypobaric hypoxia) are less prone to develop type 2 diabetes mellitus as compared to individuals living at sea-level (normobaric normoxia). Furthermore, there is evidence to suggest that normobaric hypoxia exposure may improve glucose homeostasis and insulin sensitivity in both rodents and humans.

The level of physical activity is an important determinant of insulin sensitivity and glucose homeostasis. It is well established that performing physical activity improves glucose uptake in the short term, and glycemic control in the long term. Interestingly, recent studies have demonstrated that an acute bout of exercise under hypoxic conditions (inhalation of air containing less oxygen) may lead to a more pronounced improvement in plasma glucose concentrations and/or insulin sensitivity as compared to normoxic exercise. However, the effects of repeated hypoxic exercise bouts on glucose profile throughout the day (i.e. 24h continuous glucose monitoring) remain elusive. In the present randomized, placebo-controlled, single-blind, cross-over study study, the investigators will investigate the effects of exercise under mild normobaric hypoxic conditions (FiO2, 15%) for 4 consecutive days (2 x 30-min cycling session at 50% WMAX) on postprandial substrate metabolism and 24h-glucose level in overweight/obese subjects with impaired glucose tolerance. The investigators hypothesize that 4 consecutive days of exposure to mild hypoxia while performing moderate intensity exercise improves glucose homeostasis in overweight and obese individuals with impaired glucose homeostasis.

DETAILED DESCRIPTION:
In the present randomized, single-blind, placebo-controlled cross-over study, subjects will be exposed to normobaric 1) mild hypoxia (oxygen level: 15%) and 2) normoxia (oxygen level: 21%) during exercise (2 x 30min/day on a cycle ergometer) of the same relative exercise intensity (equal to 50%WMAX under normoxic conditions) for 4 consecutive days. Subjects will be randomly assigned to each condition (computer-generated randomization plan; block size, n=4), separated by a washout period (3-6 weeks). To accomplish this, subjects will exercise in an oxygen chamber in which oxygen concentration of the ambient air and, as such, oxygen levels can be tightly controlled and monitored. Subjects will cycle two times a day for 30 minutes at 50% WMAX, determined by an incremental workload test. Since we will allow 5-10 min for subjects to get ready to start the 30-min exercise session, and take into account a 5-min cooling down period before leaving the hypoxic room again, subjects will be in the room for 45 min for each session.

After initial screening, subjects are asked to visit the university for two periods of 5 consecutive days each with a washout period of 3-6 weeks. During the first 4 days (time investment: 4.5 hours/day), subjects will be undergoing the exercise regimen, as described above.

* At day 1, on the first morning of each regimen, a glucose sensor (Enlite Glucose Sensor MiniMed; Medtronic). The sensor will be inserted subcutaneously, will be inserted subcutaneously, at 5 cm from the umbilicus, on the right side of the abdomen, and will be connected to a continuous glucose monitor (iPro2 Professional CGM MiniMed; Medtronic, Northridge, CA, USA). The sensor will remain inserted throughout the study (days 1-5). Furthermore, a physical activity monitor (ActivPAL3 micro monitor) will be applied at the same moment, to monitor physical activity of participants. At the end of day 5, the glucose sensor, and the physical activity monitor will be removed.
* At days 1-5 (time investment: 4.5 hours), fasting blood samples will be collected to determine plasma metabolites and inflammatory markers, and blood pressure and body weight will be monitored.
* At day 5 (time investment: 8 hours), a mixed liquid meal challenge will be performed to determine fasting and postprandial metabolite concentrations, and substrate oxidation (using indirect calorimetry). A skeletal muscle biopsy (m. vastus lateralis) will be collected under fasting conditions. Moreover, HOMA-IR will be used to estimate insulin resistance, using fasting plasma glucose and insulin values measured on the day after completion of the 4 day regimen.

After initial screening, the assessment of basal metabolic rate (BMR) and the incremental workload test (to determine the maximal workload, WMAX), subjects will have to invest approximately 52 hours.

ELIGIBILITY:
Inclusion Criteria:

* overweight or obese (BMI >28 kg/m2)
* impaired glucose tolerance (2h glucose: >7.8 - 11.1 mmol/L)
* subjects have to be weight-stable for at least 3 months prior to participation (no change in bodyweight: <3kg change)

Exclusion Criteria:

* cardiovascular disease (determined by questionnaire, blood pressure (Subjects with moderate to severe hypertension (grade 2 or 3 based on WHO criteria)
* type 2 diabetes mellitus
* cancer
* asthma
* bronchitis
* chronic obstructive pulmonary disease
* lung fibrosis
* obstructive sleep apnea
* use of oxygen at home situation
* resting SpO2 ≤93%
* abnormal pre-bronchodilator forced expiratory volume (FEV1) and forced vital capacity (FVC)
* liver or kidney malfunction (determined based on ALAT and creatinine levels, respectively)
* disease with a life expectancy shorter then 5 years
* lactose intolerance
* abuse of products (alcohol consumption > 15 units/week)
* smoking
* plans to lose weight (subjects will be asked if they have weight loss plans (e.g. to increase their physical activity level or change diet)
* use of high doses of anti-oxidant vitamins
* use of any medication that influences glucose metabolism and inflammation
* shift working

Ages: 30 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
Average 24 hour glucose concentration (at day 4) | Change of average glucose concentration compared to moderate intensity exercise under normoxia (21% oxygen) at day 4
  Glucose concentration will be measured in the interstitial fluid of the subcutaneous adipose tissue every 5 min using a glucose sensor (Enlite Glucose Sensor MiniMed; Medtronic) (iPro2 Professional CGM MiniMed; Medtronic, Northridge, CA, USA), which will be inserted subcutaneously, at 5 cm from the umbilicus, on the right side of the abdomen, and will be connected to a continuous glucose monitor (iPro2 Professional CGM MiniMed; Medtronic, Northridge, CA, USA). The cumulative effects of the 4 day exercise regimens will be determined using the average 24h glucose levels collected on day 4.

SECONDARY OUTCOMES:
Glycemic variability over 24 hours | Change of glycemic variability over 24 hours compared to moderate intensity exercise under normoxia (21% oxygen) at day 2, 3, 4 and 5
  Moderate intensity exercise under mild hypoxia compared to normoxia. The cumulative effects of the 4 day exercise regimens will be determined using the 24h glucose levels collected on day 4. Glycemic variability, which reflects acute glucose fluctuations, will be assessed by the standard deviation of the average 24 h glucose concentration (SD)
Time in hyper/hypoglycaemia | Change of time spent in hyper/hypoglycemia compared to moderate intensity exercise under normoxia (21% oxygen) at day 2, 3, 4 and 5
  Moderate intensity exercise under mild hypoxia compared to normoxia. The cumulative effects of the 4 day exercise regimens will be determined using the 24h glucose levels collected on day 4 frequency and duration of hypo- and hyperinsulinemia will be monitored using the iPro2 device and Enlite Glucose Sensor (Medtronic) and is defined as a glucose level of ≥10.0 mmol/l for hyperglycemia, whilst hypoglycemia will be defined as a glucose concentration ≤3.9 mmol/l.
Energy expenditure | Change of energy expenditure compared to moderate intensity exercise under normoxia (21% oxygen) at day 5 during the meal-test
  Moderate intensity exercise under mild hypoxia compared to normoxia. Energy expenditure will be determined by means of indirect calorimetry at day 5 (under normoxia in both periods), after 4 consecutive days of performing exercise under normoxia or mild hypoxia.
Substrate oxidation | Change of substrate oxidation compared to moderate intensity exercise under normoxia (21% oxygen) at day 5 during the meal-test
  Moderate intensity exercise under mild hypoxia compared to normoxia. Substrate oxidation (e.g. carbohydrate and fat oxidation) will be determined by means of indirect calorimetry at day 5 (under normoxia in both periods), after 4 consecutive days of performing exercise under normoxia or mild hypoxia.
Systolic and diastolic blood pressure | Change of systolic and diastolic blood pressure compared to moderate intensity exercise under normoxia (21% oxygen) at day 1, 2, 3, 4 and 5 under fasting conditions.
  Moderate intensity exercise under mild hypoxia compared to normoxia. Every morning, before having breakfast, systolic and diastolic blood pressure will be monitored in mmHg.
HOMA-IR | Change of HOMA-IR compared to moderate intensity exercise under normoxia (21% oxygen) at day 5 under fasting conditions
  Moderate intensity exercise under mild hypoxia compared to normoxia. HOMA-IR will be determined from circulating insulin and glucose levels at sampled at day 5.
Gene/protein expression of AMPK and phosphorylation of AMPK in skeletal muscle tissue | Change of gene/protein expression of AMPK in skeletal muscle tissue compared to moderate intensity exercise under normoxia (21% oxygen) at day 5, under fasting conditions, when skeletal muscle biopsy will be collected
  Moderate intensity exercise under mild hypoxia compared to normoxia. Skeletal muscle biopsy will be performed at day 5 under fasting conditions and will be analysed for histology and gene/protein expression. Gene expression will be performed by targeted q-PCR (quantitative-polymerase chain reaction), and protein expression will be performed by means of Western blotting to quantify expression of AMPK.
Systemic concentration of interleukin-8 (IL-8; inflammatory marker) | Change of concentrations of IL-8 compared to moderate intensity exercise under normoxia (21% oxygen) during fasting conditions at day 5
  Moderate intensity exercise under mild hypoxia compared to normoxia. At day 5, fasting blood will be sampled and analysed for systemic inflammatory markers by means of ELISA
Systemic concentration of tumor necrosis factor alpha (TNF-alpha; inflammatory marker) | Change of concentrations of TNF-alpha compared to moderate intensity exercise under normoxia (21% oxygen) during fasting conditions at day 5
  Moderate intensity exercise under mild hypoxia compared to normoxia. At day 5, fasting blood will be sampled and analysed for systemic inflammatory markers by means of ELISA
Systemic concentration of interferon-gamma (IFN-gamma; inflammatory marker) | Change of concentrations of IFN-gamma compared to moderate intensity exercise under normoxia (21% O2) during fasting conditions at day 5
  Moderate intensity exercise under mild hypoxia compared to normoxia. At day 5, fasting blood will be sampled and analysed for systemic inflammatory markers by means of ELISA
Systemic concentration of interleukin-6 (IL-6; inflammatory marker) | Change of concentrations of IL-6 compared to moderate intensity exercise under normoxia (21% oxygen) during fasting conditions at day 5
  Moderate intensity exercise under mild hypoxia compared to normoxia. At day 5, fasting blood will be sampled and analysed for systemic inflammatory markers by means of ELISA
Fasting and postprandial plasma glucose concentration | Change of fasting and postprandial plasma glucose concentrations (mmol/L) compared to moderate intensity exercise under normoxia (21% oxygen) at day 5
  Moderate intensity exercise under mild hypoxia compared to normoxia. At day 5, fasting and postprandial circulating glucose concentrations (mmol/L) will be determined during a high-carbohydrate mixed-meal test.
Fasting and postprandial plasma insulin concentration | Change of fasting and postprandial plasma insulin concentrations (mU/L) compared to moderate intensity exercise under normoxia (21% oxygen) at day 5
  Moderate intensity exercise under mild hypoxia compared to normoxia. At day 5, fasting and postprandial circulating insulin concentrations (mU/L) will be determined during a high-carbohydrate mixed-meal test.
Fasting and postprandial plasma free fatty acids concentration | Change of fasting and postprandial plasma free fatty acids concentrations (μmol/L) compared to moderate intensity exercise under normoxia (21% oxygen) at day 5
  Moderate intensity exercise under mild hypoxia compared to normoxia. At day 5, fasting and postprandial circulating free fatty acids concentrations (μmol/L) will be determined during a high-carbohydrate mixed-meal test.
Fasting and postprandial plasma glycerol concentration | Change of fasting and postprandial plasma glycerol concentrations (μmol/L) compared to moderate intensity exercise under normoxia (21% oxygen) at day 5
  Moderate intensity exercise under mild hypoxia compared to normoxia. At day 5, fasting and postprandial circulating glycerol (μmol/L) will be determined during a high-carbohydrate mixed-meal test.
Fasting and postprandial plasma triglycerides concentration | Change of fasting and postprandial plasma triglycerides concentrations (μmol/L) compared to moderate intensity exercise under normoxia (21% oxygen) at day 5
  Moderate intensity exercise under mild hypoxia compared to normoxia. At day 5, fasting and postprandial circulating triglycerides (μmol/L) will be determined during a high-carbohydrate mixed-meal test.
Fasting and postprandial plasma lactate concentration | Change of fasting and postprandial plasma lactate concentrations (mmol/L) compared to moderate intensity exercise under normoxia (21% oxygen) at day 5
  Moderate intensity exercise under mild hypoxia compared to normoxia. At day 5, fasting and postprandial circulating lactate (mmol/L) will be determined during a high-carbohydrate mixed-meal test.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Human Biology, Maastricht University Medical Centre, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No